CLINICAL TRIAL: NCT00639561
Title: Effect of Controlled Diets on Structural and Functional Dynamic of the Human Intestinal Microflora
Brief Title: Calibrated Diets and Human Intestinal Microflora
Acronym: AlimIntest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: University Hospital of Grenoble, Direction de la recherche clinique
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DCIC 06 12
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: Bacteria
Keywords: digestive system; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): diet composed of 10g of fibre per day
  Interventions: Dietary Supplement: 10 g of fibres per day
- B (Experimental): diet composed of 40g of fibre per day
  Interventions: Dietary Supplement: 40 g of fibres per day

INTERVENTIONS:
Dietary Supplement: 10 g of fibres per day — 10 g of fibres per day
  Other Names: low fibres
  Arms: A
Dietary Supplement: 40 g of fibres per day — 40g of fibres per day
  Other Names: high fibres
  Arms: B

SUMMARY:
The main objective of the study is to realized a collection of feces in order to study the modification of the intestinal microflora according to alimentary fibres

DETAILED DESCRIPTION:
Human intestinal tract count up to 1014 bacteria. We consider that each bacterial flora is composed of more than 500 different species among which only 20% are cultivable. Although this flora is well unknown, it is known that it play a major role in the metabolism of the eating fibers. Dysfunctions of this flora may be implied in numerous local and general pathologies.

It has been shown that probiotics and prebiotics are able to act upon the intestinal flora. On the basis of the personal real-life, it is generally considered acquired that our diet modifies this flora. However not many studies have validated this hypothesis with human normal diet (not artificially enriched with prebiotics or probiotics). The idea that our diet can modified the functioning of our intestinal flora (and so favor certain pathologies or activate recovery) is widely hypothetic.

A best knowledge of the diversity of this flora and to put at disposal tools to study it on a large scale could allow to answer this question. The demonstration that some food components could modify the composition or the functioning of this flora would have considerable consequences in medicine and food processing industry.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18,5 and 25

Exclusion Criteria:

* Antibiotherapy in the previous month
* Current Antibiotherapy
* Gastro-intestinal dysfunction
* Pregnancy, parturient and feeding woman
* Person deprived of freedom by judiciary or administrative decision, person in legal protection,
* Prebiotic and/or osmotic laxatives in the previous month
* Preparation for coloscopy in the previous month

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Modification of the composition or of the functioning of the intestinal microflora during calibrated diets | at day 1, 4 and 5 of each diet

SECONDARY OUTCOMES:
Modification of the composition or of the functioning of the intestinal microflora during spontaneous diets | before, between and after calibrated diets

CONTACTS AND LOCATIONS:
Overall Officials: Eric Fontaine, MDPhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Clinical research center, Grenoble, France

REFERENCES:
- [Background] Suau A, Bonnet R, Sutren M, Godon JJ, Gibson GR, Collins MD, Dore J. Direct analysis of genes encoding 16S rRNA from complex communities reveals many novel molecular species within the human gut. Appl Environ Microbiol. 1999 Nov;65(11):4799-807. doi: 10.1128/AEM.65.11.4799-4807.1999. PMID 10543789
- [Background] Aaltonen LA, Peltomaki P, Leach FS, Sistonen P, Pylkkanen L, Mecklin JP, Jarvinen H, Powell SM, Jen J, Hamilton SR, et al. Clues to the pathogenesis of familial colorectal cancer. Science. 1993 May 7;260(5109):812-6. doi: 10.1126/science.8484121.
- [Background] Moore WE, Moore LH. Intestinal floras of populations that have a high risk of colon cancer. Appl Environ Microbiol. 1995 Sep;61(9):3202-7. doi: 10.1128/aem.61.9.3202-3207.1995. PMID 7574628
- [Background] Black AE, Coward WA, Cole TJ, Prentice AM. Human energy expenditure in affluent societies: an analysis of 574 doubly-labelled water measurements. Eur J Clin Nutr. 1996 Feb;50(2):72-92. PMID 8641250
- [Background] Robinson RR, Feirtag J, Slavin JL. Effects of dietary arabinogalactan on gastrointestinal and blood parameters in healthy human subjects. J Am Coll Nutr. 2001 Aug;20(4):279-85. doi: 10.1080/07315724.2001.10719048. PMID 11506055
- [Background] Tuohy KM, Kolida S, Lustenberger AM, Gibson GR. The prebiotic effects of biscuits containing partially hydrolysed guar gum and fructo-oligosaccharides--a human volunteer study. Br J Nutr. 2001 Sep;86(3):341-8. doi: 10.1079/bjn2001394. PMID 11570986
- [Background] Chinda D, Nakaji S, Fukuda S, Sakamoto J, Shimoyama T, Nakamura T, Fujisawa T, Terada A, Sugawara K. The fermentation of different dietary fibers is associated with fecal clostridia levels in men. J Nutr. 2004 Aug;134(8):1881-6. doi: 10.1093/jn/134.8.1881. PMID 15284370